CLINICAL TRIAL: NCT02247921
Title: A Randomized Controlled Trial on Rehabilitation Through Caregiver-delivered Nurse-organized Service Programs for Disabled Stroke Patients in Rural China
Brief Title: Rehabilitation for Disabled Stroke Patients in Rural China
Acronym: RECOVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute for Global Health, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CMB13-161
Record Dates: First submitted 2014-09-13; First posted 2014-09-25 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Stroke
Keywords: caregiver delivered rehabilitation; nurse-organized service; disabled stroke patients
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rehabilitation (Experimental): nurse-led caregiver-delivered rehabilitation
  Interventions: Other: Rehabilitation
- Usual care (No Intervention): The patients in the control arm will receive conventional care in terms of access to rehabilitation in hospital, timeliness of discharge and follow-up, without any explicit provision of caregiver training or accelerated discharge.

INTERVENTIONS:
Other: Rehabilitation — Patients recruited into the intervention arm will have their family-nominated caregivers trained by a trained nurse and guided by a culturally appropriate and easy-to-understand rehabilitation manual to be given to caregivers at the last session, shortly before hospital discharge to reduce contamination. The training sessions will take at least 90 minutes per day for 2 or 3 days.The nurse will call the patients and caregivers at 2, 4, and 8 weeks after hospital discharge to monitor progress and offer guidance on rehabilitation.Duration of the standardized yet individualized intervention by nurses will be 8 weeks; however, trained caregivers are expected to deliver the rehabilitation services to patients as long as they are needed.
  Arms: Rehabilitation

SUMMARY:
Stroke is the second leading cause of mortality and disability among adults worldwide. Rehabilitation is an effective treatment for stroke; however rehabilitation services are far from adequate in China, especially in rural areas where the health and economic burden of disability from stroke is very high.

The investigators propose to develop, implement, and evaluate an evidence-based caregiver-delivered stroke rehabilitation program designed to improve the physical functioning of disabled stroke patients in rural China.

DETAILED DESCRIPTION:
This randomized controlled trial will be conducted in Zhangwu People's Hospital in Liaoning Province, Qingtongxia People's Hospital in Ningxia Hui Autonomous Region and Dianjiang People's Hospital in Chongqing City. Eligible and consenting stroke in patients with residual disability will be randomized into the intervention group or control group after they have passed the acute care stage and approved by their physicians to be recruited into the study. Standardized baseline assessments for all patients include Barthel Index (activities of daily living), modified Rankin Scale, and other demographic, disease history, lifestyle, and health information. Nurses in the county hospital will be trained by rehabilitation specialists and will in turn train the family caregivers of patients in the intervention group with the aid of an easy-to-understand picture-rich rehabilitation manual, specially designed for this study. The content of training is based on 10 domains in the Barthel Index, which can be classified into 3 groups: mobility, self-care, and toileting. Nurses will do the telephone based follow-up to patients at approximately 2, 4, and 8 weeks post-discharge to provide follow-up care and consultation. Follow-up evaluation of all patients will be conducted by researchers not involved in the intervention. Pre-discharge evaluation including Barthel Index, modified Rankin Scale and Functional Ambulation Category will be conducted face to face with patients, . 3 months and 6 months evaluation will be conducted via telephone based interview.3 months evaluation includes living condition, Barthel Index ,modified Rankin Scale, hospitalization condition and medicine usage. Based on 3 months evaluation, 6 months evaluation includes additional measures: Functional Ambulation Classification, EQ-5D, 9-item Patient Health Questionnaire, physical examination and caregiver burden. Primary outcome will be the Barthel Index score at 6-month after hospital discharge. The study will be conducted in 2 phases: 1) pilot study (Lasting for 2 months, 30 patients in Zhangwu People's Hospital and 30 patients in Qingtongxia People's hospital); and 2) main study (Lasting for 15 months, 100 patients in Zhangwu People's Hospital, 100 patients in Qingtongxia People's hospital and 60 patients in Dianjiang People's Hospital). Information from pilot study will be used for refinement of the intervention and study implementation. Patients in the pilot study will be followed until the end of the study, resulting in a total of 320 patients.

Primary Hypothesis: The innovative caregiver-delivered nurse-organized rehabilitation intervention, compared to usual care, will significantly improve physical functioning of disabled stroke patients in rural China, as measured by the Barthel Index (activities of daily living) at six months after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years，and≤79 years);
* Recent (<1 month) first-ever acute ischemic/hemorrhagic/undifferentiated stroke patients;or recurrent patients with the result of Modified Rankin Scale (MRS) no more than 2 points.
* With a reasonable expectation of 6 month survival post-discharge (i.e. not palliative, no evidence of widespread cancer etc.);
* Residual disability (requiring physical assistance for core activities of daily living defined as a Barthel Index score of 80 or lower)

Exclusion Criteria:

* Unable to identify a suitable family-nominated caregiver for training and subsequent delivery of care
* Unable to provide informed consent from both the patient (or by proxy) and the caregiver

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2014-08; Primary Completion 2016-12-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Barthel Index (activities of daily living) at 6 months | 6 months

SECONDARY OUTCOMES:
Barthel Index at 3 months | 3 months
Functional Ambulation Classification (FAC) at 6 months | 6 months
EQ-5D quality of life at 6 months | 6 months
Patient Health Questionnaire - 9 items at 6 months | 6 months
Modified Rankin Scale at 3 and 6 months | 3 and 6 months

OTHER OUTCOMES:
Caregiver Burden Index at 6 months | 6 months
hospitalization | 6 months
medical costs | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lijing Yan, Principal Investigator — Duke Kunshan University
Locations (1):
- The Georgeinstitute of Global Health at Peking University Health Science Center, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhou B, Zhang J, Zhao Y, Li X, Anderson CS, Xie B, Wang N, Zhang Y, Tang X, Prvu Bettger J, Chen S, Gu W, Luo R, Zhao Q, Li X, Sun Z, Lindley RI, Lamb SE, Wu Y, Shi J, Yan LL. Caregiver-Delivered Stroke Rehabilitation in Rural China. Stroke. 2019 Jul;50(7):1825-1830. doi: 10.1161/STROKEAHA.118.021558. Epub 2019 Jun 10. PMID 31177978